CLINICAL TRIAL: NCT05831215
Title: Development and Validation of the Italian Version of the Modified Barthel Index and of the Motricity Index Scales
Brief Title: Italian Version of the Modified Barthel Index
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Other Study IDs: mBI - MI - part B
Record Dates: First submitted 2023-02-03; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2022-12

CONDITIONS: Cross-Cultural Comparison; Validation Study; Reliability and Validity; Disability Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to develop and validate the Italian version of the modified Barthel Index (mBI-Italian), through the following steps:

* translation of the mBI into Italian, by using the froward-backward translation approach, to produce a pre-final mBI-Italian
* pre-pilot testing of the pre-final mBI-Italian in a sample of ten health professionals (physicians and physiotherapists), ten subjects who had a stroke, and 10 caregivers, i.e. subjects who take care of a person who had a stroke. All participants will be asked to judge the clarity of each item of the scale, including scoring instructions
* evaluation of the metric properties (internal consistency, inter- and intra-rater reliability, validity and responsiveness) of the final mBI-Italian in a sample of subjects admitted to the Don Gnocchi Foundation in Florence for rehabilitation after stroke

DETAILED DESCRIPTION:
The modified Barthel Index (mBI) (Shah et al (1989) is a worldwide adopted scale which investigates independence in the basic activities of daily living. It comprises ten items as the original version (personal hygiene, bathing, feeding, toilet, stairs, dressing, bowels, bladder, transfers, ambulation/wheelchair management), with a modification to the scoring to enhance its responsiveness. The mBI has been cross-culturally adapted in several countries and languages, However, despite unofficial versions circulating in clinical settings, there is currently no validated Italian version of the scale. This study aims to develop this version and to evaluate its metric properties in a sample of subjects who had a stroke.

A pre-final mBI-Italian will be produced following established international guidelines (forward-backward translation, each step involving two different translators). This version will be tested in a group of ten health professionals (physicians and physiotherapists), ten subjects who had a stroke and ten caregivers, All participants will be asked to judge the clarity of each item of the scale, including scoring instructions, using a dichotomous response (clear/unclear). Items that are judged unclear by more than 20 percent of evaluators will be revised by the multidisciplinary translation team to produce the final mBI-Italian.

The final mBI-Italian will then be administered to a sample of at least 100 subjects with stroke to assess its metric properties in this population. Participants will be enrolled among patients admitted to the Don Gnocchi Foundation in Florence for stroke rehabilitation. To assess reliability, upon admission each patient will be independently assessed using the mBI-Italian by two examiners, drawn at random from a group of ten physiotherapists. One of the two raters will administer the scale twice on consecutive days. Other evaluators will administer other clinical scales (Fugl-Meyer assessment, FMA; modified Rankin scale, mRS) to assess the validity of the mBI-Italian. All raters will be blinded to all other assessments and to their previous assessment, if any. All the scales will be administered again at discharge, when participants will also be asked to indicate the perceived change since admission in their ability to autonomously manage the basic activities of daily living (ADLs). For the latter, a 7-points Global Rating of Perceived Change (GRPC) Lickert scale will be used.

The Cronbach's alpha will be used to estimate the internal consistency of the scale. To assess intra-rater and inter-rater reliability, the Intraclass Correlation Coefficient (ICC1,1), Standard Error of the Measurement (SEM) and Minimal Detectable Change with 95% Confidence (MDC95) will be computed. Criterion and construct validity will be assessed by computing the association between the mBI-Italian and the FMA and the mRS, at both admission and discharge. For responsiveness, the following indices will be calculated: 1) Guyatt Responsiveness Index (GRI); 2) Standardized Response Mean (SMR), both in the whole sample and in subgroups of participants with different outcome (improved, unchanged, worsened) based on the GPRC; 3) Minimal Clinically Important Difference (MCID). The latter will be derived using the ROC curve approach, using the patient's perceived change in his/her autonomy in basic ADLs as an anchor.

ELIGIBILITY:
The study is divided in two phases: A) pilot-testing of the pre-final mBI-Italian, and B) verification of the metric properties (reliability, validity and responsiveness) of the final mBI-Italian.

A) Pilot-test of the pre-final mBI-Italian (verification of clarity of all items):

Inclusion criteria:

Health professionals:

* Being a physician or a physiotherapist with at least three
* years of experience in the functional assessment of subjects with stroke;
* willingness to participate in the study.

Subjects who had a stroke:

* age 18 years or older
* stroke outcomes such that they impact the person's ability to independently perform various basic activities of daily living
* willingness to participate in the study, with informed consent signed (by the support administrator/legal guardian, if necessary)

Caregivers:

* age 18 years or older;
* Being a person who takes care of a disabled subject who had a stroke;
* willingness to participate in the study,

Exclusion criteria:

Health professionals: none

Subjects who had a stroke:

* severe visual and/or auditory impairment that cannot be corrected
* cognitive impairment defined by a Mini Mental State Examination (MMSE) score <21;
* severe language impairment such that comprehension and performance of the task is prevented
* presence of signs of clinical instability, defined by a score greater than zero on the Clinical Instability Scale

Caregivers:

* severe visual and/or auditory impairment that cannot be corrected
* cognitive impairment defined by a Mini Mental State Examination (MMSE) score <21
* severe language impairment such that comprehension and performance of the task is prevented.

B) Study on the metric properties of the final mBI-Italian:

1. Participants (subjects who had a stroke): all patients consecutively admitted to the Don Gnocchi Foundation of Florence for rehabilitation after stroke (until the expected sample size is completed) who meet the following criteria.

   Inclusion criteria:
   * age 18 years or older
   * stroke outcomes such that they impact the person's
   * ability to independently perform various basic activities of daily living
   * willingness to participate in the study, with informed consent signed (by the support administrator/legal guardian, if necessary)

   Exclusion criteria:
   * severe visual and/or auditory impairment that cannot be corrected
   * cognitive impairment defined by a Mini Mental State Examination (MMSE) score <21
   * severe language impairment such that comprehension and performance of the task is prevented
   * presence of signs of clinical instability, defined by a score greater than zero on the Clinical Instability Scale
2. Raters: ten physiotherapists with at least three years of experience in the evaluation and treatment of subjects with stroke outcomes. Pairs of raters, equal in number to the number of patients enrolled, will be randomly drawn from this group, and each pair will be randomly assigned to a patient to be administered the mBI-IT. Other examiners, also randomly drawn from the list of ten raters, will administer other clinical scales to participants to assess the validity of the mBI-IT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A) In the pilot-testing, the pre-final versione of the mBI-Italian will be tested for clarity on a sample of 10 health professionals (physicians and physiotherapists) working in stroke rehabilitation, 10 subjects who had a stroke and 10 caregivers.
  B) The metric properties of the final mBI-italian will be tested on a sample of at least 100 patients who had a stroke. Considering a possible dropout rate of 15 percent, 115 subjects are expected to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Internal Consistency - Baseline assessment | Assessment at admission (T0).
  Cronbach's alpha
Internal Consistency - Discharge assessment | Assessment at discharge (T1). Time of discharge will vary among participants, so a definite time point cannot be stated. On average, discharge is expected after about 30 days from admission.
  Cronbach's alpha
Intra-rater reliability | Test and Retest assessments, conducted 1-3 days apart.
  One-way random-effects model sIngle measures Intraclass Correlation Coefficient (ICC1,1).
Inter-rater reliability | Assessment at admission conducted independently by two independent raters 30-60 minutes apart.
  One-way random-effects model sIngle measures Intraclass Correlation Coefficient (ICC1,1).
Intra-rater reliability (error of measurement) | Test and Retest assessments, conducted 1-3 days apart.
  Standard Error of the Measurements (SEM), computed as the standard deviation of the two measures collected by the same rater, multiplied by the square root of 1 minus ICC.
Inter-rater reliability (error of measurement) | Assessment at admission conducted independently by two independent raters 30-60 minutes apart.
  Standard Error of the Measurements (SEM), computed as the standard deviation of the measures collected by two independent raters, multiplied by the square root of 1 minus ICC.
Intra-rater reliability (Minimal Detectable Change) | Test and Retest assessments, conducted 1-3 days apart.
  Minimal Detectable Change at the 95 % confidence level (MDC 95), computed as the SEM multiplied by 1,96 multiplied by the square root of 2.
Inter-rater reliability (Minimal Detectable Change) | Assessment at admission conducted independently by two independent raters 30-60 minutes apart.
  Minimal Detectable Change at the 95 % confidence level (MDC 95), computed as the SEM multiplied by 1,96 multiplied by the square root of 2.
Criterion Validity - Association with reference standard at admission. | Assessment at admission (T0).
  Estimation of the correlation between the mBI-Italian and the modified Rankin Scale (mRS).
Criterion validity - Association with reference standard at discharge. | Assessment at discharge (T1). Time of discharge will vary among participants, so a definite time point cannot be stated. On average, discharge is expected after about 30 days from admission.
  Estimation of the correlation between the mBI-Italian and the mRS.
Construct validity (hypothesis testing) - Association with sensorimotor impairment at admission. | Assessment at admission (T0).
  Estimation of the correlation between the mBI-Italian and the Fugl-Meyer Assessment (FMA) scale.
Construct validity (hypothesis testing) - Association with sensorimotor impairment at discharge. | Assessment at discharge (T1). Time of discharge will vary among participants, so a definite time point cannot be stated. On average, discharge is expected after about 30 days from admission.
  Estimation of the correlation between the mBI-Italian and the FMA scale.
Responsiveness (change of mBI scores from admission to discharge) - Standardized Response Mean (SRM). | Admission (T0) and Discharge (T1) assessment. Time of discharge will vary among participants, so a definite time point cannot be stated. On average, discharge is expected after about 30 days from admission.
  For each subject, the change score at the mBI-Italian will be calculated as the difference between T1 and T0 assessment. The SRM will be calculated as the ratio of observed change and the standard deviation reflecting the variability of the change scores, both in the whole sample and separately in groups with different outcome based on the Global Rating of Perceived Change (GRPC).
Responsiveness (change of mBI scores from admission to discharge) - Guyatt Responsiveness Index (GRI). | Admission (T0) and Discharge (T1) assessment. Time of discharge will vary among participants, so a definite time point cannot be stated. On average, discharge is expected after about 30 days from admission.
  For each subject, the change score at the mBI-Italian will be calculated as the difference between T1 and T0 assessment. The GRI will be calculated as the ratio of the mean change score difference between improved and stable patients and the standard deviation of the individual change scores in stable patients. Improved and stable patients will be detected based on the GRPC.
Responsiveness (change of mBI-Italian scores from admission to discharge) - Minimal Clinically Important Difference (MCID). | Admission (T0) and Discharge (T1) assessment. Time of discharge will vary among participants, so a definite time point cannot be stated. On average, discharge is expected after about 30 days from admission.
  For each subject, the change score at the mBI-Italian will be calculated as the difference between T1 and T0 assessment. The Receiving Operator Characteristic (ROC) curve approach will be used to estimate the minimal change score associated with clinically important change (i.e., the MCID), using the GRPC as an anchor.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Cecchi F, Cassio A, Lavezzi S, Scarponi F, Gatta G, Montis A, Bernucci C, Franceschini M, Bargellesi S, Paolucci S, Taricco M. Redefining a minimal assessment protocol for stroke rehabilitation: the new "Protocollo di Minima per l'ICtus" (PMIC2020). Eur J Phys Rehabil Med. 2021 Oct;57(5):669-676. doi: 10.23736/S1973-9087.21.06638-7. Epub 2021 May 27. PMID 34042407
- [Background] MAHONEY FI, BARTHEL DW. FUNCTIONAL EVALUATION: THE BARTHEL INDEX. Md State Med J. 1965 Feb;14:61-5. No abstract available. PMID 14258950
- [Background] Shah S, Vanclay F, Cooper B. Improving the sensitivity of the Barthel Index for stroke rehabilitation. J Clin Epidemiol. 1989;42(8):703-9. doi: 10.1016/0895-4356(89)90065-6. PMID 2760661
- [Background] Sousa VD, Rojjanasrirat W. Translation, adaptation and validation of instruments or scales for use in cross-cultural health care research: a clear and user-friendly guideline. J Eval Clin Pract. 2011 Apr;17(2):268-74. doi: 10.1111/j.1365-2753.2010.01434.x. Epub 2010 Sep 28. PMID 20874835